CLINICAL TRIAL: NCT01235156
Title: A Single-dose, Open Labeled, Multicenter Phase IIa Clinical Study on the Efficacy and Safety of Sulcardine Sulfate Tablets in Patients With Premature Ventricular Contractions
Brief Title: Efficacy and Safety of Sulcardine Sulfate Tablets in Patients With Premature Ventricular Contractions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiangsu Furui Pharmaceuticals Co., Ltd (Industry)
Responsible Party: A Single-dose, Open labeled, Multicenter Phase IIa Clinical Study on the Efficacy and Safety of Sulcardine Sulfate Tablets in Patients with Premature Ventricular Contractions, Jiangsu Furui Pharmaceuticals Co., Ltd
Other Study IDs: TG0823SUL
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-11

CONDITIONS: Premature Ventricular Contraction
Keywords: Premature ventricular contraction; Frequent premature ventricular contraction, with or without a short array of non-sustained ventricular tachycardia
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Arrhythmia is a common disease that may be caused by various cardiovascular diseases. According to statistics, 500,000 people die of severe arrhythmia every year in China, In the United States, approximately 540,000 patients die each year.This study will evaluate the effectiveness safety of sulcardine sulfate tablets in the patients with premature ventricular contractions (and non-sustained VT).

DETAILED DESCRIPTION:
Arrhythmia is a common disease that may be caused by various cardiovascular diseases. The incident rate of various types of arrhythmias may be as high as 86-100% in patients who experience acute myocardial infarction within 10 days. Serious arrhythmias can endanger lives instantly. According to statistics, 500,000 people die of severe arrhythmia every year in China, which constitutes approximately 50% of the death rate for cardiovascular diseases. In the United States, among 1,500,000 myocardial infarction patients, approximately 540,000 patients die each year, which is mainly caused by ventricular fibrillation (VF) and sudden cardiac death (SCD).

Initially at least 24 subjects who meet the inclusion criteria and do not meet the exclusion criteria will be enrolled into either of two dose levels under a 3:1 randomization (active:placebo) take sulcardine sulfate tablets.Dose levels may be dropped, an intermediate dose level added as needed to deemed appropriate following review of safety and tolerability data at the prior dose level(200mg,400mg). A safety review committee will review data from all enrolled subjects at the simultaneous completion of Dosing Cohort 1 and 2 prior to advancement to the final dose level (800mg BID).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, body weight 45-80kg, and no sex preference.
2. Frequent premature ventricular contraction, the total number of premature ventricular beats indicated by Holter monitor greater than 3600 over 24 hours, with or without a short array of non-sustained ventricular tachycardia (more than 3, but fewer than 10 consecutive ventricular beats).
3. Negative pregnancy test result within 24 hours before the first dose for women of childbearing age. Females subjects of child bearing age must be on effective birth control (IUD or compliant use of oral contraceptive), have been surgically sterilized or abstain from sexual intercourse through the active dosing period and for the first 10 days after dosing.
4. Voluntary participation in the study and the ability to complete the screening and trial procedures, and to remain in the clinical study site throughout dosing period in accordance with the protocol.
5. Understand and voluntarily sign a written informed consent document.

Exclusion Criteria:

1. History of Stage III-IV congestive heart failure.
2. Ejection fraction <35% predicted
3. Polymorphic ventricular tachycardia, sustained ventricular tachycardia.
4. Congenital or acquired long QT syndrome, Torsade de Pointes, or an uncorrected QT-interval of >480 ms; QRS>120 ms.
5. Unstable angina, active myocarditis, rheumatic fever, or bacterial endocarditis, elevated Troponin T on work-up.
6. Sinus node dysfunction, atrioventricular block above first degree not controlled by pacemaker.
7. Complete left or right bundle branch block, or intraventricular block.
8. Hypotension, sitting resting blood pressure below 90/55mmHg.
9. Hypertension as defined by SBP> 160mmHg and/or DBP > 95mmHg
10. Sinus bradycardia (average heart rate lower than 50 beats/min).
11. Liver (liver function tests or bilirubin (direct or indirect) >2XULN, history of cirrhosis or chronic active hepatitis.
12. Kidney dysfunction (plasma creatinine>1.8 and creatinine clearance calculation <30 as determined by Cockroft-Gault calculation) or electrolyte or acid-base balance disorders.
13. Taking digitalis, tricyclic antidepressants, β blockers, or calcium channel blockers within 5 half-lives for a given agent.
14. Thyroid dysfunction.
15. Serious respiratory diseases, Wolff-Parkinson-White syndrome; chronic obstructive pulmonary disease, asthma requiring medication
16. Cyanotic or other uncorrected significant congenital heart disease.
17. History of allergy to sulfonamides.
18. Taking other anti-arrhythmic drugs or medications that affect cardiac electrophysiology, or stop taking the above mentioned medications less than 5 half-life of the drug ago.
19. History of taking amiodarone within 1 years.
20. Severe neurosis, menopausal syndrome, chest pain caused by cervical spondylosis.
21. Diseases of the hematopoietic system, or mental illness.
22. Current evidence of alcohol abuse or history of illegal drug abuse.
23. Women of childbearing potential who are pregnant or nursing, or women of childbearing age who are not on effective birth control (IUD or compliant use of oral contraceptives and who have a positive urine pregnancy test prior to study.
24. Participation in a clinical trial of other drugs within 3 months.
25. Those considered not suitable to be selected by the investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-70 year-old patients with premature ventricular contractions or non-sustained ventricular tachycardia (VT)
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2010-11

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing chao-yang hosipital, Beijing, Beijing Municipality
  - Peking university people's hosipital, Beijing, Beijing Municipality